CLINICAL TRIAL: NCT03794063
Title: Analysis of Caesarean Section Rate According to the 10 Group Robson Classification; A Multicenter Prospective Study in Egypt
Brief Title: Analysis of Caesarean Section Rate According to the Robson Classification System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Egyptian Society of Royal College of Obstetricians and Gynaecologists (Other)
Responsible Party: Principal Investigator, Dr Bismeen Jadoon, Research coordinator, Egyptian Society of Royal College of Obstetricians and Gynaecologists
Other Study IDs: ERC-RCOG
Record Dates: First submitted 2018-12-29; First posted 2019-01-04 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Caesarean Section Rate
Keywords: Robson classification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Robson group 1: Nulliparous women, single cephalic, more than or equal to 37 weeks, in spontaneous labour
  Interventions: Other: Robson 10 group classification system
- Robson Group 2: Nulliparous women, single cephalic, more than or equal to 37 weeks, induced or Caesarean section before labour
  Interventions: Other: Robson 10 group classification system
- Robson Group 3: Multiparous women with out a previous Caesarean section , with a single cephalic pregnancy, more than or equal 37 weeks gestation in spontaneous labour
  Interventions: Other: Robson 10 group classification system
- Robson Group 4: Multiparous women with out a previous Caesarean section , with a single cephalic pregnancy, more or equal 37 weeks gestation who had labour induced or were delivered by Caesarean section before labour
  Interventions: Other: Robson 10 group classification system
- Robson Group 5: All Multiparous women with at least one CS with a single cephalic pregnancy, more or equal to 37 weeks gestation
  Interventions: Other: Robson 10 group classification system
- Robson Group 6: All nulliparous women with a single breech pregnancy
  Interventions: Other: Robson 10 group classification system
- Robson Group 7: Multiparous women with a single breech pregnancy including women with previous Caesarean section
  Interventions: Other: Robson 10 group classification system
- Robson Group 8: All women with multiple pregnancies including women with previous Caesarean sections
  Interventions: Other: Robson 10 group classification system
- Robson Group 9: All women with a single pregnancy with a transverse or oblique lie, including women with previous Caesarean Section (s)
  Interventions: Other: Robson 10 group classification system
- Robson Group 10: All women with a single cephalic pregnancy less than 37 weeks gestation, including women with previous Caesarean section (s)
  Interventions: Other: Robson 10 group classification system

INTERVENTIONS:
Other: Robson 10 group classification system — WHO proposed the Robson classification system as a global standard for assessing, monitoring and comparing caesarean section rates within healthcare facilities over time, and between facilities. It classifies women in 10 groups based on their obstetric characteristics (parity, previous CS, gestational age, onset of labour, fetal presentation and number of fetuses) without needing the indication for CS.

SUMMARY:
A prospective cross- sectional study will be conducted to implement the Robson Classification to assess, analyze and compare Caesarean section rate of the participating hospital over the period of three months. The Robson implementation manual will be used as a tool guide for the study.

DETAILED DESCRIPTION:
Increase rate of unnecessary caesarean sections has been a growing concern in most parts of the world. According to the latest survey one in five women in the world now deliver by caesarean section (CS). The Eastern Mediterranean Region (EMR) with its twenty -two Member States (MSs) as classified by the World Health Organization is of no exception in this respect. Within the EMR, Egypt has the highest CS rate of 54%, with no further improvement to maternal and child mortality rates in Egypt, the association of extremely high CS rate and its potential benefits has been questioned. This may suggest that although the necessary numbers of CSs are performed for the population at risk but the rates higher than the recommended threshold (10-15% according to the WHO) could be the measure of unjustified CSs in healthy populations . However, determining the adequate caesarean section rate at the population level - i.e. the minimum rate for medically indicated caesarean section, while avoiding medically unnecessary operations - is a challenging task. Variations in overall CS rate between different settings or over time are difficult to interpret and compare because of intrinsic differences in hospital factors and infrastructure (primary versus tertiary level), difference in the characteristics of the obstetric population (case mix) served (eg % of women delivered by previous CS) and difference in clinical management protocols. This is seen as one of the barriers in better understanding of CS trends and underlying causes. In order to propose and implement effective measures to achieve optimal CS rates, it is first essential to identify what groups of women are contributing the most towards overall CS rate and investigate the underlying reasons for trends in different settings. Like many developing countries, health care facilities in Egypt have no such standardized internationally accepted classification system in place to monitor and compare facility based CS rates in a consistent and action oriented manner.

Policy makers and health organisations have suggested the need for such classification system that can best monitor and compare CS rates in a standardised, reliable, consistent and action-oriented manner. WHO proposed the Robson classification system as a global standard for assessing, monitoring and comparing caesarean section rates within healthcare facilities over time, and between facilities. It classifies women in 10 groups based on their obstetric characteristics (parity, previous CS, gestational age, onset of labour, fetal presentation and number of fetuses) without needing the indication for CS. It gives an opportunity to evaluate the prevalence of CSs among various groups of women, to compare data between institutions, learn from each other and to create strategies for better results through audit and feed back cycle. This classification is clinically relevant and categorizes women prospectively which in turns allows the implementation and evaluation of interventions targeted to specific groups. Some studies have shown that if this classification is used on a regular basis, it can provide critical assessment to change the practice.

Aim: The study aim is, to assess, analyse and compare CSR of the participating hospital over the period of three months according to the 10 Group Robson classification system

Participating hospitals

1: Ain Shams University Hospital 4: Mataria Teaching Hospital 4: Shatby Alexandria Hospital 5: Benha University Hospital 6: Ahmed Maher Hospital 7: El-Galaa Hospital 8: Alexandria Hospital 9: Behira Hospital 10:Menia Hospital 11: Luxor Hospital 12: Nada Hospital 13: Rofayda Hospital

Study design: A prospective cross- sectional study will be conducted to implement the Robson Classification within the obstetric department of participating hospitals. The Robson implementation manual will be used as a tool guide for the study.

The study population will include all women with live births and stillbirths of at least 28 weeks gestation at from. Two-study investigator from each participating hospital will be assigned who will provide the ongoing support during the study period. Participants will be invited to attend the introductory workshop for the implementation of the Robson Classification by the study coordinators. Variables necessary to categorise women in to Robson groups will be collected through the predesigned proforma. These variables will be used to classify each woman in to Robson groups with the help of a flow diagram. The collected information will be analyzed on the Excel Sheet to finalize the grouping either manually or by an automatic calculator.The results of each group will be statistically analyzed after entering the data in the report and will be sent on a monthly basis by e-mail or fax to study coordinators.

ELIGIBILITY:
Inclusion criteria:

* Women delivering at ≥ 28 weeks gestation

Exclusion Criteria:

* Women delivering at < 28 weeks gestation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women admitted to the labour ward for delivery who are 28 or more weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
caesarean section rate | three months
  absolute and relative caesarean section rate

SECONDARY OUTCOMES:
Postpartum haemorrhage | from 24 hours to 6 weeks after the delievry
  1. Blood loss of more than 500 mls at vaginal birth
  2. Blood loss of more than 1000 mls at caesarean section
Maternal morbidity | 7 days after the delivery
  Admission to Intensive care unit after the delivery
Neonatal morbidity | 7 days of the delivery
  Admission of newborn to Neonatal intensive care unit
Maternal mortality | 42 days after the delivery
  maternal death from 24 hours to 42 days after the delivery
Neonatal mortality | 28 days after the delivery
  death during the first 28 days of life (0-27 days

CONTACTS AND LOCATIONS:
Locations (1):
- Egyption society of Royal college of obstetricians and gynaecologist, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months after the study completed

REFERENCES:
- [Background] Appropriate technology for birth. Lancet. 1985 Aug 24;2(8452):436-7. PMID 2863457
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Torloni MR, Betran AP, Souza JP, Widmer M, Allen T, Gulmezoglu M, Merialdi M. Classifications for cesarean section: a systematic review. PLoS One. 2011 Jan 20;6(1):e14566. doi: 10.1371/journal.pone.0014566. PMID 21283801
- [Background] Betran AP, Vindevoghel N, Souza JP, Gulmezoglu AM, Torloni MR. A systematic review of the Robson classification for caesarean section: what works, doesn't work and how to improve it. PLoS One. 2014 Jun 3;9(6):e97769. doi: 10.1371/journal.pone.0097769. eCollection 2014. PMID 24892928
- [Background] Robson MS (2001) Classification of caesarean sections. Fetal and Maternal Medicine Review 12: 23-39.
- [Background] Robson M, Hartigan L, Murphy M. Methods of achieving and maintaining an appropriate caesarean section rate. Best Pract Res Clin Obstet Gynaecol. 2013 Apr;27(2):297-308. doi: 10.1016/j.bpobgyn.2012.09.004. Epub 2012 Nov 3. PMID 23127896
- [Background] Boatin AA, Cullinane F, Torloni MR, Betran AP. Audit and feedback using the Robson classification to reduce caesarean section rates: a systematic review. BJOG. 2018 Jan;125(1):36-42. doi: 10.1111/1471-0528.14774. Epub 2017 Jul 17. PMID 28602031
- [Background] Chaillet N, Dumont A. Evidence-based strategies for reducing cesarean section rates: a meta-analysis. Birth. 2007 Mar;34(1):53-64. doi: 10.1111/j.1523-536X.2006.00146.x. PMID 17324180
- See also: Egypt Demographic Health Survey (DHS) , 2014 — http://dhsprogram.com/pubs/pdf/FR302/FR302.pdf